CLINICAL TRIAL: NCT04342910
Title: A Study of Camrelizumab (SHR-1210) Combined With Apatinib Versus Paclitaxel or Irinotecan in Participants With Advanced Gastric/Gastroesophageal Junction Adenocarcinoma Progressed After First-line Chemotherapy
Brief Title: Study to Evaluate the Efficacy and Safety of Camrelizumab and Apatinib in Patients With GC/GEJC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR-1210-III-316
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; apatinib; Paclitaxel; Irinotecan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- camrelizumab (SHR-1210) combined with apatinib (Experimental): Participants will receive camrelizumab on Day 1 and Day 15 of each 28-day cycle and apatinib mg/day up to 2 years.
  Interventions: Drug: camrelizumab; Drug: Apatinib Mesylate
- Paclitaxel or Irinotecan (Active Comparator): Participants receive paclitaxel on Days 1, 8, and 15 of each 28-day cycle, or irinotecan on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Paclitaxel; Drug: Irinotecan

INTERVENTIONS:
Drug: camrelizumab — 200 mg intravenous (IV) camrelizumab on Day 1 and Day 15 of each 28-day cycle.
  Other Names: SHR-1210
  Arms: camrelizumab (SHR-1210) combined with apatinib
Drug: Apatinib Mesylate — 250 mg qd
  Arms: camrelizumab (SHR-1210) combined with apatinib
Drug: Paclitaxel — 80 mg/m^2 administered as IV infusion on Days 1, 8, and 15 of each 28-day cycle.
  Arms: Paclitaxel or Irinotecan
Drug: Irinotecan — 180 mg/m^2 administered as IV infusion on Days 1, and 15 of each 28-day cycle.
  Arms: Paclitaxel or Irinotecan

SUMMARY:
This is a study for participants with advanced gastric or gastroesophageal junction adenocarcinoma who have had tumor progression after first-line platinum-contained therapy. The primary study hypotheses are that camrelizumab (SHR-1210) combined with apatinib prolongs overall survival (OS) for participants with tumors that show positive programmed cell death ligand 1 (PD-L1) expression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- or cytologically-confirmed diagnosis of gastric or gastroesophageal junction adenocarcinoma.
2. Confirmed metastatic or locally advanced, unresectable disease.
3. Progression on or after prior first-line therapy containing any platinum/fluoropyrimidine or platinum/taxane doublet.
4. Willing to provide tumor tissue for PD-L1 biomarker analysis.
5. Human epidermal growth factor receptor 2 (HER-2/neu) status known and participants with HER2/neu positive tumors show documentation of previous treatment containing trastuzumab.
6. ECOG performance status of 0 to 1.
7. Life expectancy of more than 12 weeks.
8. Signing the informed consent forms.
9. Adequate bone marrow, liver and renal function.

Exclusion Criteria:

1. Squamous cell or undifferentiated gastric cancer.
2. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. Subjects with an active, known or suspected autoimmune disease. Patients with type I diabetes who are receiving a stable dose of insulin, hypothyroidism who only needs hormone replacement therapy, and skin diseases (such as eczema, vitiligo, or psoriasis) that do not require systemic treatment and do not have acute deterioration within 1 year before the screening period, are allowed.
4. Clinically significant cardiovascular and cerebrovascular diseases.
5. Subjects with high blood pressure who cannot be controlled well with antihypertensive drugs.
6. Previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency.
7. Arterial / venous thrombosis events, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism, occurred within the first 6 months of randomization.
8. Subjects who have previously received anti-PD-1 / PD-L1 monoclonal antibody, anti-CTLA-4 monoclonal antibody, and VEGFR small molecule inhibitor therapy.
9. Prior systemic chemotherapy, radiotherapy and surgery within 4 weeks before the study drug administration, or any unresolved AEs > Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in PD-L1 Positive Participants. | Up to 27 months
  OS was defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) in All Participants. | Up to 27 months
  OS was defined as the time from randomization to death due to any cause.
Progression-free Survival (PFS) According to RECIST 1.1 base on investigator assessment in All Participants or in PD-L1 Positive Participants. | Up to 27 months
  PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator assessment, or death due to any cause, whichever occurs first.
Time to Tumor Progression (TTP) According to RECIST 1.1 based on investigator assessment in All Participants or in PD-L1 Positive Participants. | Up to 27 months
  TTP was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator assessment in All Participants.
Time to Failure (TTF) in All Participants or in PD-L1 Positive Participants | Up to 27 months
  TTF was defined as the time from randomization to treatment discontinuation caused by any reason.
Objective Response Rate (ORR) According to RECIST 1.1 based on investigator assessment in All Participants or in PD-L1 Positive Participants. | Up to 27 months
  ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR or PR according to RECIST 1.1 based on investigator assessment.
Duration of Response (DOR) According to RECIST 1.1 Based on investigator assessment in All Participants or in PD-L1 Positive Participants. | Up to 27 months
  DOR was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) According to RECIST 1.1 based on investigator assessment in All Participants or in PD-L1 Positive Participants. | Up to 27 months
  DCR was defined as the percentage of the participants in the analysis population who had a confirmed CR or PR or SD according to RECIST 1.1 based on investigator assessment.
Time to Response (TTR) According to RECIST 1.1 based on investigator assessment in All Participants or in PD-L1 Positive Participants. | Up to 27 months
  TTR was defined as the time from randomization to the first documented evidence of CR or PR.
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v4.03. | Up to 27 months
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) as assessed by CTCAE v4.03.
Proportion of dose suspension, dose reduction or dose discontinuation caused by treatment-related toxicities. | Up to 27 months
  Proportion of dose suspension, dose reduction or dose discontinuation caused by treatment-related toxicities.
Proportion of anti-camrelizumab antibody (ADA) and neutralizing antibody (Nab) formed during the study from baseline | Up to 27 months
  Proportion of anti-camrelizumab antibody (ADA) and neutralizing antibody (Nab) formed during the study from baseline
Serum concentration of camrelizumab | Up to 27 months
  Serum concentration of camrelizumab
Plasma concentration of apatinib | Up to 27 months
  plasma concentration of apatinib

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Ph.D, Principal Investigator — Affiliated Hospital, Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital, Academy of Military Medical Sciences, Beijing, China